CLINICAL TRIAL: NCT04285710
Title: Adjunctive Phototherapy Treatment of Infected Diabetic Ulcers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was never started since the IRB application was not submitted and the PI left the institution.
Sponsor: Boston Medical Center (Other)
Collaborators: Ji-Xin Cheng Laboratory (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-38602
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Diabetic Foot; Diabetic Foot Ulcer; Diabetes; Diabetes Mellitus; Infected Wound; Infected Ulcer of Skin
Keywords: Phototherapy; Blue Light Phototherapy; Light Therapy
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Wound Infection | interventions — Phototherapy; Bandages; Debridement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (Other): Subjects enrolled in the subject group will receive standard care treatment for infected diabetic wounds, including debridement surgery and wound dressings. However, in order to maintain consistency with the phototherapy arm, subjects within the control group will visit the clinic twice a week, with the first visit being for the debridement surgery, and the second visit being for clinical wound dressing redressing.
  Interventions: Procedure: Debridement Surgery and Wound Dressing
- Phototherapy (Experimental): For this intervention therapy, subjects enrolled in the experimental group will still receive standard care treatment for infected diabetic wounds. However, experiment group subjects will receive phototherapy treatments alongside standard care. A mobile pulsed laser device will be utilized to apply nanosecond pulsed 410 nm light onto both the cellulitis afflicted regions and open wound portions of a patient's infected diabetic ulcer wound twice a week over the course of the 3 month study. The device will be designed and produced by the Ji Xin Cheng Lab located at the Boston University Charles River Campus. Phototherapy sessions will occur twice a week, with the first session occurring after debridement surgery, and the second session occurring later in the week during clinical wound dressing redressing.
  Interventions: Device: Phototherapy; Procedure: Debridement Surgery and Wound Dressing

INTERVENTIONS:
Device: Phototherapy — The key intervention aspect of this study is the application of 15 J/cm2 of 410 nm pulsed light directly onto the infected diabetic wounds of subjects every week over the course of 3 months, allowing for the cumulative exposure of around 180 J/cm2 for the entire study. This 15 J/cm2 weekly dosage of blue light will split up into two sessions every week, with each session applying 7.5 J/cm2 of light treatment. Phototherapy will be applied twice per week, with one phototherapy session occurring directly following the debridement surgery during the first visit of the week and the other session occurring after the study clinician removes the subjects wound dressings at the second visit.
  Other Names: OPOTEK Opolette HE 355 LD Tunable Laser
  Arms: Phototherapy
Procedure: Debridement Surgery and Wound Dressing — All patients enrolled in the study will undergo standard care and treatment for infected diabetic wounds, which includes the weekly surgical removal of infected necrotic tissue from the diabetic wounds. In addition to debridement, both groups will utilize an antimicrobial wound dressing to cover and treat the infected diabetic wound. The subject's wounds will be dressed with Aquacel Ag Advantage Wound Dressings to protect and treat their diabetic wounds. These dressings will be changed twice a week by clinicians.
  Other Names: Debridement

SUMMARY:
The key purpose of this study is to determine and understand the safety and effectiveness of blue light phototherapy in the treatment and healing of infected diabetic wounds, as well as determining if this treatment is capable of reducing the bacterial population number within infected wounds. The investigators' lab recently discovered that a specific survival protein called catalase can be destroyed through blue light exposure. Given that a majority of bacteria species contains catalase, it is hypothesized that the destruction of this protein can improve the effectiveness of antimicrobial wound dressings commonly used to treat infected diabetic wounds, therefore further reducing the amount of bacteria within the wound and increasing the rate of healing. By reducing the overall bacterial population within these diabetic infected wounds, the ability for these diabetic wounds to heal will be enhanced, allowing for greater reductions in wound size over the course of the treatment.

In this study, 40 subjects will be enrolled and randomly assigning subjects to either a control group or a phototherapy receiving experimental group. While control subjects will receive standard weekly debridement treatment procedures for infected diabetic ulcers, experimental subjects will receive standard weekly debridement treatment alongside 2 sessions of phototherapy every week over the course of 12 weeks. Bacterial swab samples will be taken alongside the excised debrided infect tissue for the purpose of bacterial population analysis. For each patient, the changes in total bacterial population, wound size, and subject satisfaction will be recorded and analyzed to determine the effectiveness of pulsed light phototherapy.

ELIGIBILITY:
Inclusion Criteria:

* English Speaking
* Capacity to Consent
* Diabetic Foot Ulcers
* Have an infected wound present on the foot greater than 1 (one) cm2 and less than 8 cm2
* Ability to utilize appropriate offloading devices as recommended by a clinician

Exclusion Criteria:

* Pregnant or breastfeeding/nursing
* Ankle-brachial pressure index below 0.45 or over 1.4
* Hemoglobin A1c levels above 12.0
* Stage 4 renal disease/dialysis
* Taking immunosuppressant medications
* Undergoing radiation therapy
* Diagnosed Uncontrolled/Resistant hypertension (HTN) - High blood pressure that does not respond well to medical treatment, blood pressure remains above average (usually 130/80 mmHg) despite medication usage.
* Diagnosed Uncontrolled malabsorption disorder - Small intestine unable to absorb nutrients effectively, usage of nutrient supplements ineffective
* Active sepsis
* Uncontrolled coagulopathy - Blood unable to properly coagulate and form clots, low platelet or clotting factor levels, unresponsive to medications
* Untreated bone/soft tissue infection - Not yet initially treated to reduce risk of sepsis
* Gangrene of wound under care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Bacterial Quantification Over Time | 12 weeks
  Bacterial swabs will be collected from each subject's wound before and after weekly debridement. These weekly bacterial swabs, in addition to the homogenized debrided tissue, will be used to assess a patient's overall bacterial burden and bacterial population. Overall bacterial counts and population within each sample will be determined through the use of colony-forming unit (CFU) counting on agar plates or bacterial sequencing.

SECONDARY OUTCOMES:
Wound Size Reduction Over Time | 12 weeks
  Participants will have their diabetic wounds imaged and measured on a week-to-week basis, determining the changes in wound area and cellulitis afflicted area.
Subject Phototherapy Treatment Satisfaction: questionnaire | 12 weeks
  An investigator developed questionnaires will be completed each week by the participants that asks questions about their overall satisfaction with the treatment regimen and whether changes will need to be made to the phototherapy treatment procedure to ensure a better patient experience.

CONTACTS AND LOCATIONS:
Overall Officials: David Negron, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No